CLINICAL TRIAL: NCT04678479
Title: Expanded Access With Adjunctive Ganaxolone Treatment in Children and Young Adults With Cyclin Dependent Kinase-like 5 Deficiency Disorder
Brief Title: Ganaxolone Expanded Access Program Compassionate Use
Acronym: CDD
Status: No longer available | Type: Expanded Access
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 1042-CDD-EAP-3005
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: CDKL5 Disorder
MeSH Terms: conditions — CDKL5 deficiency disorder | interventions — ganaxolone

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Drug: Ganaxolone — ganaxolone

SUMMARY:
The primary objective is to provide GNX to patients ≥ 2 years with CDD-related seizures who are refractory to, or intolerant of, standard therapy.

DETAILED DESCRIPTION:
This is a multi-center, long-term, open-label, expanded access protocol of adjunctive GNX treatment in children, adolescents, and adults with CDD. Patients with inadequate seizure control on their current anti seizure medications at therapeutic doses will be eligible for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Molecular confirmation of a pathogenic CDKL5 variant, early onset, difficult to control seizures, and neurodevelopmental impairment are required. Male or female patients aged ≥ 2 years. In the opinion of the investigator, the patient has inadequate seizure control on current anti-seizure medications at therapeutic doses.

Exclusion Criteria:

-

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Paula Bokesch, MD, FAAP, Study Director — Marinus Pharmaceuticals, Inc.; Igor Grachev, MD, PhD, Study Director — Marinus Pharmaceuticals, Inc.